CLINICAL TRIAL: NCT06389890
Title: Pancreatic Surgery - Optimal Caseload Thresholds and Predictive Accuracy
Acronym: PaSuT
Status: Completed | Type: Observational
Sponsor: Richard Hunger (Other)
Collaborators: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Sponsor-Investigator, Richard Hunger, Principal Investigator, Medizinische Hochschule Brandenburg Theodor Fontane
Organization: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Other Study IDs: PaSuTE
Record Dates: First submitted 2024-03-15; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Volume-Outcome Relationship in Pancreatic Surgery
Keywords: Outcome Assessment; General Surgery; Pancreatic Surgery; Public Health; Hospital Planning; Centralized Hospital Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- All patients undergoing pancreatic surgery: All patients with at least one pancreatic surgery procedure code
  Interventions: Procedure: Pancreatic resection procedure
- Subgroup: Total pancreatectomy: All patients with at least one of the following pancreatic procedure codes (OPS-codes): '55250', '55251', '55252', '5525x', '5525y'
  Interventions: Procedure: Pancreatic resection procedure
- Subgroup: Pancreaticoduodenectomy: All patients with at least one of the following pancreatic procedure codes (OPS-codes): '55241', '55242', '55243'
  Interventions: Procedure: Pancreatic resection procedure
- Subgroup: Segmental resection: All patients with at least one of the following pancreatic procedure code (OPS-codes): '55244'
  Interventions: Procedure: Pancreatic resection procedure
- Subgroup: Distal pancreatectomy: All patients with at least one of the following pancreatic procedure codes (OPS-codes): '55240', '552400', '552401', '552402'
  Interventions: Procedure: Pancreatic resection procedure
- Subgroup: Other partial resections: All patients with at least one of the following pancreatic procedure codes (OPS-codes): '5524x', '5524y'
  Interventions: Procedure: Pancreatic resection procedure

INTERVENTIONS:
Procedure: Pancreatic resection procedure — Pancreatic resection procedure

SUMMARY:
The main objective of the study is to identify the optimal annual number of cases in a hospital with regard to minimising hospital mortality in pancreatic surgery. In particular, the prognostic value of such case numbers will be analysed.

DETAILED DESCRIPTION:
Main research questions:

* Can specific intervention case numbers be identified that are suitable as thresholds for annual minimum volumes and are associated with significantly low hospital mortality?
* Almost all previous studies on case number effects have only shown a descriptive association between the number of cases in a given year and the quality of outcomes in the same year. The aim of this study is to investigate whether the correlations described can be demonstrated when using the previous year's procedure volume as a predictor. The study seeks to answer whether the procedure caseload has predictive value, specifically the number of cases in one year and in-hospital mortality in the following year.

Background:

Numerous studies have demonstrated a correlation between the number of cases and the quality of outcomes for various surgical procedures. For instance, patients who underwent surgery in high-volume hospitals (HVH) had lower mortality rates, longer survival rates, lower complication rates, and lower reoperation rates than patients who underwent surgery in low-volume hospitals (LVH). To subdivide into HVHs and LVHs, either concrete case numbers or quartile or quintile limits with an equal number of operations or clinics per group wer used. The aim of the study is to objectively determine these limits using a spline-modeled caseload term, avoiding arbitrary decisions.

One limitation of the previous findings is that they may not be generalisable due to the use of a limited number of cases and outcome quality from the same year. However, it is important to note that the volume from the previous year is crucial in determining the predictive importance of caseload for future outcome quality. A recent study (in press) reported, that there are significant fluctuations in the quality of outcomes among HVHs, even between different years. Therefore, it was hypothesized that using the number of cases as a predictor of high-quality outcomes may lead to overestimation.

Methods:

The nationwide hospital billing data for Germany (DRG statistics) for the period 2010 to 2019 will be analysed. The risk-adjusted mortality rates are determined. For this purpose, logistic regression models are calculated that adjust the mortality risk for the following variables Sex, age, emergency of admission, year of resection, diagnosis (malign neoplasm vs. benign neoplasm vs. neoplasm of unclear dignity vs. acute pancreatitis vs. chronic pancreatitis vs. other pancreatic diseases), additional procedures (venous resections/ multivisceral resections/ arterial resections/ splenectomy/ cholecystectomy/ biliary drainage/ dialysis procedures) and selected comorbidities. To classify additional procedures in order to reflect extent of surgery and technical difficulty, a slight modification of the classification system as described in Mihaljevic et al, 2021 will be used (PMID: 33386130). The Elixhauser definitions are used for the comorbidities as described in Quan et al, 2005 (PMID: 16224307). The selection of comorbidities to be considered is based on the publication by Hunger et al, 2022 (PMID: 35525416).

The case number effect is modelled using natural cubic splines. The 10th, 20th, 40th, 60th, 80th and 90th case number percentiles are used as node points. The adjusted hospital mortality as a function of the number of cases is determined using Estimated Marginal Means. Local extremes (maxima and minima) in the splines are determined using 1st and 2nd graph derivate.

Various regression models are calculated using either the number of cases from the current year of operation or the previous year. The predictive accuracy of the models is determined using the established measures from signal detection theory (AUC, sensitivity, specificity, positive predictive value, negative predictive value). Subgroup analyses for individual resection procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* any pancreatic resection procedure
* operated at any German hospital

Exclusion Criteria:

* any transplantation procedure
* Inpatient admission for organ removal
* no information on sex
* no information on age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population encompasses all patients that underwent any pancreatic resection procedure in any German hospital (full survey of the German population).
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | within 30 days
  Patient died during or after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rene Mantke, MD, Study Director — Head of Surgery at University Hospital Brandenburg an der Havel

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed by controlled remote data analysis. The data is held exclusively by the Federal Statistical Office for scientific analyses. Direct access to or data sharing of individual patient data is prohibited by German law.